CLINICAL TRIAL: NCT00923351
Title: A Pilot Study of Tumor Vaccination and R-hIL-7 Following Standard Multimodality Therapy in Patients With High Risk Pediatric Solid Tumors
Brief Title: Therapy to Treat Ewing's Sarcoma, Rhabdomyosarcoma or Neuroblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Glod, Staff Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070206; 07-C-0206; NCT00526240 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Neuroblastoma; Sarcoma; Rhabdomyosarcoma-Embryonal; Rhabdomyosarcoma- Alveolar; Neuroectodermal Tumors, Primitive, Peripheral
Keywords: Vaccine; Immunotherapy; Cancer; Chemotherapy; Tumor Lysate/KLH Pulsed Dendritic Cell Vaccine; Neuroblastoma; Autologous Lymphocyte Infusion; Ewing's Sarcoma; Rhabdomyosarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Rhabdomyosarcoma, Embryonal; Rhabdomyosarcoma, Alveolar; Neuroectodermal Tumors, Primitive, Peripheral; Neoplasms; Sarcoma, Ewing; Rhabdomyosarcoma | interventions — efineptakin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Participants who did not receive rhIL-7 (Experimental): Six patients with Ewings sarcoma family or tumors (ESFT) participants will receive cytotoxic/lympholytic therapy with cyclophosphamide and fludarabine (if cluster of differentiation 4 (CD4) count > 200 cells/mcl). Participant will receive Tumor lysate/keyhole limpet hemocyanin (KLH) pulsed dendritic cell vaccine followed by Infusion of 8H9/CD25 depleted autologous lymphocyte infusion on Day 1, followed by Tumor lysate/KLH pulsed dendritic cell vaccine on week 4, 6, 8, 10, and 12.
  Interventions: Drug: Tumor Purged/CD25 Depleted Lymphocytes
- Arm B - Participants who received rhIL-7 (Experimental): Eight patients with rhabdomyosarcoma, fifteen patients with Ewings sarcoma family or tumors (ESFT), two patients with desmoplastic small round cell tumor, and one patient with synovial cell sarcoma participants will receive CYT107 20 mcg/kg/dose subcutaneous (SQ) (approx. 48h prior to vaccine[Day 0]), Tumor lysate/KLH pulsed dendritic cell vaccine followed by Infuse 8H9/CD25 depleted autologous lymphocyte infusion on Day 2, followed by CYT107 20 mcg/kg/dose SQ on days 14, 28 and 42 (± 7 days), and Tumor lysate/KLH pulsed dendritic cell vaccine on Days 16, 30, 44, 56, and 70 (± 7 days).
  Apheresis/flow cytometry/delayed type of hypersensitivity (DTH) responses for immune endpoint monitoring (skin tests) will be performed on Week 8, 14, 20 (Arm A) and on Days 42, 84 and 126 (+/- 7 days) (Arm B); and radiographic studies for clinical restaging will be performed on Week 8 and 20 (Arm A) and Days 42 and 126 (+/- 7 days) (Arm B).
  Interventions: Biological: Tumor Purged/CD25 Depleted Lymphocytes with Tumor Lysate/KLH Pulsed Dendritic Cell Vaccine; Drug: rhIL-7; Biological: Tumor Lysate/KLH Pulsed Dendritic Cell Vaccine

INTERVENTIONS:
Drug: Tumor Purged/CD25 Depleted Lymphocytes
  Arms: Arm A - Participants who did not receive rhIL-7
Biological: Tumor Purged/CD25 Depleted Lymphocytes with Tumor Lysate/KLH Pulsed Dendritic Cell Vaccine — Tumor lysate/KLH pulsed dendritic cells (minimum of 1 X 10e6 cells/kg) on Day2.
  Arms: Arm B - Participants who received rhIL-7
Drug: rhIL-7 — rhIL-7 (20 mcg/kg/dose SQ) approx. 48 hours prior to vaccine) Day 0, Day 14, Day 28 and Day 42
  Arms: Arm B - Participants who received rhIL-7
Biological: Tumor Lysate/KLH Pulsed Dendritic Cell Vaccine — Tumor lysate/KLH Pulsed dendritic cell vaccine (1-5 X 10e7 cells/injection site, given in 3 sites intradermal) on Day 2, Day 16, Day 30, Day 44, Day 56, Day 70.
  Arms: Arm B - Participants who received rhIL-7

SUMMARY:
Background:

* Pediatric solid tumors (Ewing's sarcoma, rhabdomyosarcoma, and neuroblastoma) are often difficult to cure with standard treatment.
* Immune therapy using an experimental vaccine made from proteins from the patient's tumor cells may boost the body's immune response against the tumor.
* The effects of chemotherapy on the immune system can potentially make immunotherapy more effective if administered soon after completion of chemotherapy. The addition of recombinant human IL-7 (interleukin 7) (rhIL-7 (recombinant human interleukin 7)) may make the immunotherapy more effective.

Objectives:

-To determine whether immune therapy given after immune suppression can help the body fight the tumor and to determine the safety of the treatment.

Eligibility:

-Patients with solid tumors, i.e., Ewing's sarcoma, rhabdomyosarcoma or neuroblastoma whose disease has recurred after treatment or spread beyond the original site

Design:

* Patients undergo tumor biopsy (removal of a piece of tumor tissue) to collect tumor cells for making a vaccine from proteins in the patient's tumor and apheresis (removal of a quantity of white blood cells) to collect white cells for re-building the immune system after immune therapy. Apheresis is repeated three times during immunotherapy (weeks 8, 14 and 20).
* After receiving standard chemotherapy for their tumor (and an additional course of fludarabine and cyclophosphamide to further suppress immunity if needed) patients receive immune therapy in Cohorts A and B. rhIL-7 is given 48 hours before the vaccine, as an injection under the skin in an extremity that will not be used for the vaccine in patients in Cohort B only. You will be watched closely for 6 hours after the rhIL-7 for any signs of reaction. rhIL-7 will be given before vaccine doses #1, #2, #3, and #4. The vaccine is given at study weeks 2, 4, 6, 8, 10 and 12. Each vaccine is given as a total of six separate rhIL-7 followed by injections: three intradermal (like a (tuberculosis) TB test) on one arm or leg and three subcutaneous (like those for insulin injections for diabetes). on the other arm or leg. An anesthetic cream may be used to minimize the discomfort of injections.
* Patients' white cells are returned to them by infusion through a vein on the first day of immune therapy.
* Imaging studies and immune studies are done at weeks 1, 8 and 20 to determine the response to treatment on the tumor and on the immune system.

DETAILED DESCRIPTION:
Background:

* Patients with recurrent or metastatic pediatric solid tumors experience low survival rates, but using current standard therapies, many patients with these diseases are rendered into a state of minimal residual disease associated with lymphopenia.
* Lymphopenic hosts show augmented immune reactivity, which may be favorable for inducing antitumor immune responses.

Objectives:

* To determine whether Alpha cluster of differentiation 25 (CD25) and 8H9 depleted autologous lymphocytes plus tumor lysate/keyhole limpet hemocyanin (KLH) pulsed dendritic cell vaccines plus or minus r-hIL7 (CYT107) can induce immune responses to tumor lysate in this patient population rendered lymphopenic by cytotoxic therapy.
* To assess the safety of administering lymphocytes depleted of cluster of differentiation 4 (CD4) plus CD25plus suppressor T cells plus or minus r-hIL (CYT107 (interleukin 7)) to lymphopenic hosts.

Eligibility:

* Patients with metastatic or recurrent pediatric solid tumors of the following histologies: Ewing's sarcoma family of tumors, rhabdomyosarcoma or neuroblastoma, synovial cell sarcoma, desmoplastic small round cell tumor, undifferentiated sarcoma, embryonal sarcoma.
* Patients must have sufficient accessible tumor for biopsy to generate tumor lysate.
* Patients must meet eligibility criteria upon enrollment and upon completion of standard therapy prior to administration of immunotherapy as significant time will have elapsed between the time points.

Design:

* Immunotherapy consists of one autologous lymphocyte infusion depleted of CD25plus suppressive T cells and depleted of contaminating tumor cells plus 6 sequential tumor lysate/KLH pulsed dendritic cell vaccines. No cytokine is administered on Arm A and r-hIL7 (CYT107) is administered on Arm B.
* Patients will be evaluated for immune responses to tumor lysates using ex vivo assays and delayed type hypersensitivity (DTH).
* The trial uses a one-stage design targeting a response rate of 50 percent. Up to 47 patients will be treated.
* Stopping rules will take effect if excessive toxicity is observed.

ELIGIBILITY:
* INCLUSION CRITERIA: for Apheresis/Tumor biopsy portion of the trial:

A. Diagnosis

* rhabdomyosarcoma: embryonal or alveolar.
* Ewing's sarcoma family of tumors (ESFT), which include: classical, atypical and extraosseous ESFT, peripheral primitive neuroectodermal tumors, peripheral neuroepithelioma, primitive sarcoma of bone, and ectomesenchymoma.
* neuroblastoma: may be diagnosed via histology or the standard clinical evidence for increased catecholamines in the urine plus tumor cells in the bone marrow.
* undifferentiated or embryonal sarcoma.
* desmoplastic small round cell tumor.
* synovial cell sarcoma.

B. Extent of Disease/Previous Therapy

* Initial presentation: Stage IV or metastatic disease, enrolled prior to any cytoreductive therapy.
* Recurrent Disease:

  * Patient > 5yo must have recovered CD4 count to > 350 cells/mm^3 OR have disease free interval > one year from completion of cytotoxic therapy
  * Patients < 5yo must have recovered CD4 count to > 350 cells/mm^3 OR have disease free interval > six months from completion of cytotoxic therapy
* Multiple recurrences are allowable as long as CD4 count or disease-free intervals have been met.

C. Age/Weight

* greater than 18 mos. and less than or equal to 35 years at the time of initial diagnosis.
* greater than 10 kg at the time of apheresis. Patients between 10-15 kg must be approved by the apheresis unit prior to enrollment on protocol.

D. Informed Consent

All patients or their legal guardians (if the patient is less than 18 years old) must sign a document of informed consent (screening protocol) prior to performing studies to determine patient eligibility. After confirmation of patient eligibility all patients or their legal guardians must sign the protocol specific informed consent to document their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (other than the studies which were performed to determine patient eligibility).

E. Laboratory Parameters

* renal function: creatinine clearance greater than 60 mL/min/1.73m^2 or normal age adjusted serum creatinine (less than or equal to 5 yrs. less than or equal to 0.8 mg/ml; 5-10 yrs. less than or equal to 1.0 mg/ml; 10-15 yrs. less than or equal to 1.2 mg/ml; greater than 15 yrs. less than or equal to 1.5 mg/ml)
* liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of normal (ULN), bilirubin less than 1.5 ULN
* hematologic function: platelets greater than 50,000 cells/mcl, hemoglobin (Hgb) greater than 9.0 gms/dl, prothrombin time (PT) less than 1.5 ULN. Patients may receive transfusion if necessary to reach the pre-apheresis hematology parameters.

F. Accessibility of Tissue to Generate Tumor Lysates

Patients must have adequate tumor bulk accessible to biopsy in order to generate the tumor lysate (at least 2 cm diameter). Procedures employed to acquire biopsies for tumor lysates will be limited to percutaneous biopsies or open biopsies of readily accessible lesions. Patients should not undergo biopsies, which will later compromise the ability to render function preserving local therapy (e.g. limb salvage therapy). To prevent this, all bone biopsies should be performed in consultation with the orthopedic consultant on the case. For patients with bone marrow involvement, bone marrow aspirates may be used as a source of tumor for tumor lysates. Patients are not eligible if, in the opinion of the principal and associate investigators, tumor biopsy would entail extensive surgery such as thoracotomy or laparotomy, or if the tumor site places the patient at substantial risk from the biopsy procedure.

National Cancer Institute (NCI) Laboratory of Pathology will review all tumor specimens for diagnosis.

EXCLUSION CRITERIA: for Apheresis/Tumor biopsy portion of the trial:

A. Other conditions

* Clinically significant unrelated systemic illness, such as serious infections, autoimmunity or organ dysfunction, which in the judgment of the Principal or Associate Investigators would compromise the patient's ability to tolerate the investigational agents or are likely to interfere with the study procedures or results.
* Previous allogeneic stem cell or allogeneic bone marrow transplantation.
* Conditions related to tumor, which require emergency treatment (airway compression, spinal cord compression) since enrollment would delay initiation of such therapy.
* Women who are pregnant or lactating.
* Corticosteroids initiated at the time of tumor diagnosis or recurrence for treatment of nerve compression or other symptoms is permitted during this phase of the trial, but will not be permitted during the immunotherapy phase, with the exception of a self limited course of steroids as described in Section 2.1.4.A.
* Patients with a history of central nervous system (CNS) metastases from cancer are not excluded provided that the metastatic CNS disease has been effectively treated and there is no evidence of active CNS disease as evidenced by stable clinical findings and stable radiographic findings for a period of 6 weeks.
* Patients with human immunodeficiency virus infection, hepatitis B, or hepatitis C due to confounding effects on immune system.

INCLUSION CRITERIA: for Immunotherapy portion of the trial:

A. Informed Consent

Because significant time will have elapsed between apheresis/tumor biopsy and the initiation of immunotherapy, all patients or their legal guardians (if the patient is less than 18 years old) must sign a second informed consent to document their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (other than the studies which were performed to determine patient eligibility).

B. Time and Recovery from Cytotoxic Therapy

At least 3 weeks should have elapsed since the last cycle of cytotoxic therapy or since the last dose of radiation therapy, at least 4 weeks must have elapsed since the patient has received any investigational therapy, and patients should have recovered from toxic side effects of previous therapy to a grade 1 or less, with the exception of the following:

* Hematological toxicity: recovery to levels required in Section 2.1.1.E.
* Low electrolyte levels (Such individuals should receive appropriate supplementation).
* For patients on anticoagulant therapy or with pre-existing coagulation abnormalities, prothrombin time (PT), partial thromboplastin time (PTT) must return to baseline.
* Liver function tests must resolve to values required in Section 2.1.1.E.
* Grade 3 hypoalbuminemia.
* Alopecia.
* Sterility.

C. Laboratory Parameters

* renal function: creatinine clearance greater than 60 mL/min/1.73m^2 or normal age adjusted serum creatinine (less than or equal to 5 yrs. less than or equal to 0.8 mg/ml; 5-10 yrs. less than or equal to 1.0 mg/ml; 10-15 yrs. less than or equal to 1.2 mg/ml; greater than 15 yrs. less than or equal to 1.5 mg/ml).
* liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of normal (ULN), bilirubin less than 1.5 ULN.
* hematologic function: absolute neutrophil count (ANC) greater than 750 cells/mcl, platelets greater than 50,000 cells/mcl.

D. Birth Control

Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

EXCLUSION CRITERIA: for Immunotherapy Portion of the Trial:

A. Other conditions

* Clinically significant unrelated systemic illness, such as serious infections or organ dysfunction, which in the judgment of the Principal or Associate Investigators would compromise the patient's ability to tolerate the investigational agents or are likely to interfere with the study procedures or results.
* Persistent or progressive cancer following the completion of the standard therapy phase of the trial will not, in and of itself, preclude receipt of immunotherapy. However, patients will not receive immunotherapy if they have an Eastern Cooperative Oncology Group (ECOG) performance status performance status of 3 or 4 or, for children less than or equal to 10 years of age, Lansky less than or equal to 50 (Appendix III). Furthermore, patients will be removed from the trial if they develop requirements for anti-neoplastic therapy (e.g. radiation therapy) for progressive disease during the trial as discussed in protocol.
* Women who are pregnant or lactating.
* Patients with human immunodeficiency virus infection, hepatitis B, or hepatitis C infection due to confounding effects on immune function.
* Patients who require chronic daily oral corticosteroid or other immunosuppressive therapy. Topical or inhaled corticosteroids are permitted. Also, a time limited course of steroids does for an unrelated medical condition (e.g. allergic reaction, poison ivy) will not preclude receipt of immunotherapy provided that two weeks elapse between the last dose of systemic corticosteroids and initiation of immunotherapy.
* Patients who are receiving other biologic therapies including cytokines or growth factors not specified by the protocol. Herbal supplements will not result in exclusion but should be noted and reviewed with the principal investigator (PI).
* Patients with a history of CNS metastases from cancer are not excluded provided that the metastatic CNS disease has been effectively treated and there is no evidence of active CNS disease as evidenced by stable clinical findings and stable radiographic findings for a period of 6 weeks.
* Excluded from Arm B:

  * Patients with history of autoimmune disease (excluding thyroiditis on chronic thyroid replacement therapy) or active auto-immune disease, due to a risk of exacerbation of autoimmunity with r-hIL7. Patients with a history of B cell malignancy due to a risk for growth with rhIL7 therapy.
  * Corrected QT interval (QTc) prolongation defined as a QTc greater than or equal to 470 ms or a prior history of cardiovascular disease, arrhythmias, or significant electrocardiogram (ECG) abnormalities.

Ages: 19 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2007-06-02 (Actual); Primary Completion 2012-08-30 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arndt CA, Crist WM. Common musculoskeletal tumors of childhood and adolescence. N Engl J Med. 1999 Jul 29;341(5):342-52. doi: 10.1056/NEJM199907293410507. No abstract available. PMID 10423470
- [Background] La TH, Meyers PA, Wexler LH, Alektiar KM, Healey JH, Laquaglia MP, Boland PJ, Wolden SL. Radiation therapy for Ewing's sarcoma: results from Memorial Sloan-Kettering in the modern era. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):544-50. doi: 10.1016/j.ijrobp.2005.07.299. Epub 2005 Sep 28. PMID 16198063
- [Background] Barker LM, Pendergrass TW, Sanders JE, Hawkins DS. Survival after recurrence of Ewing's sarcoma family of tumors. J Clin Oncol. 2005 Jul 1;23(19):4354-62. doi: 10.1200/JCO.2005.05.105. Epub 2005 Mar 21. PMID 15781881
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0206.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-four patients were enrolled. Twelve patients were not treated in Arm A or B because they did not get far enough in the study to be designated for an Arm.
Groups:
- Enrolled But Not Assigned to Treatment: Twelve participants were not treated in Arm A or Arm B because they did not get far enough in the study to be designated for an Arm. Were unable to obtain apheresis, and adequate tumor samples.
Period: Overall Study
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7 | Enrolled But Not Assigned to Treatment
Started | 6 | 26 | 12
Completed | 6 | 26 | 0
Not Completed | 0 | 0 | 12
Not completed — no apheresis/adequate tumor sample | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Arm A - Participants Who Did Not Receive rhIL-7: Six patients with Ewings sarcoma family or tumors (ESFT) participants will receive cytotoxic/lympholytic therapy with cyclophosphamide and fludarabine (if cluster of differentiation 4 (CD4) count > 200 cells/mcl). Participants will receive Tumor lysate/KLH pulsed dendritic cell vaccine followed by Infusion of 8H9/CD25 depleted autologous lymphocyte infusion on Day 1, followed by Tumor lysate/KLH pulsed dendritic cell vaccine on week 4, 6, 8, 10, and 12.
- Arm B - Participants Who Received rhIL-7: Eight patients with rhabdomyosarcoma, fifteen patients with Ewings sarcoma family or tumors (ESFT), two patients with desmoplastic small round cell tumor, and one patient with synovial cell sarcoma participants will receive CYT107 20 mcg/kg/dose SQ (approx. 48h prior to vaccine[Day 0]), Tumor lysate/KLH pulsed dendritic cell vaccine followed by Infuse 8H9/CD25 depleted autologous lymphocyte infusion on Day 2, followed by CYT107 20 mcg/kg/dose SQ on days 14, 28 and 42 (± 7 days), and Tumor lysate/KLH pulsed dendritic cell vaccine on Days 16, 30, 44, 56, and 70 (± 7 days).
  Apheresis/flow cytometry/delayed type of hypersensitivity (DTH) responses for immune endpoint monitoring (skin tests) will be performed on Week 8, 14, 20 (Arm A) and on Days 42, 84 and 126 (+/- 7 days) (Arm B); and radiographic studies for clinical restaging will be performed on Week 8 and 20 (Arm A) and Days 42 and 126 (+/- 7 days) (Arm B).
- Total: Total of all reporting groups
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7 | Total
Number analyzed (Participants) | 6 | 26 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 15 | 19
  Between 18 and 65 years | 2 | 11 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (7.56) | 20.96 (8.19) | 21.0 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 20 | 22
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 20 | 26
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White (non-Hispanic) | 6 | 20 | 26
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 26 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Immune Response as Evidenced by the Delayed Type of Hypersensitivity (DTH) Reaction Assay
Description: A positive response to the tumor vaccine requires a positive reaction in at least one of the two assays below (immune responses to tumor lysates using ex vivo and delayed type of hypersensitivity (DTH).
  The presence of a positive delayed type of hypersensitivity (DTH) reaction to the tumor lysate in a patient who did not show a positive DTH reaction prior to immunotherapy. A positive reaction is induration of at least 0.5 cm.
  Immunotherapy administered to patients with recurrent or metastatic pediatric solid tumors such as Ewing's sarcoma, rhabdomyosarcoma, or neuroblastoma. Each vaccine is given as 6 separate injections. Three intradermal on one arm or leg and three subcutaneous on the other arm or leg.
Time Frame: Week 8, 14, 20 (Arm A) and on Days 42, 84 and 126 (± 7 days) (Arm B)
Population: Five of the original six participants from Arm A were analyzed because one subject was changed to a special exemption.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7
Number analyzed (Participants) | 5 | 26
Participants | 0 | 15
Statistical Analysis 1: Comparison: Arm A - Participants Who Did Not Receive rhIL-7 vs Arm B - Participants Who Received rhIL-7; Test type: Superiority or Other; p = 0.043, Fisher Exact

2. Primary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 49.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7
Number analyzed (Participants) | 6 | 26
Participants | 6 | 24

3. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time between the first day of treatment to the day of death.
Time Frame: Time between the first day of treatment to the day of death or at the conclusion of 5 years of follow-up, whichever comes first, assessed up to approximately 11 years.
Measure: Median (Full Range); unit: years
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7
Number analyzed (Participants) | 6 | 26
years | 2.4 [1.0 to 3.3] | 4.3 [0.9 to 10.4]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 49.5 months.
Arm/Group | Arm A - Participants Who Did Not Receive rhIL-7 | Arm B - Participants Who Received rhIL-7
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/26
Serious Adverse Events (participants affected / at risk) | 6/6 | 12/26
Other Adverse Events (participants affected / at risk) | 6/6 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Participants Who Did Not Receive rhIL-7 (N=6) | Arm B - Participants Who Received rhIL-7 (N=26)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 5 (5)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Infection with unknown ANC: Upper airway NOS (Infections and infestations) | 0 (0) | 1 (1)
Mood alteration: depression (Nervous system disorders) | 1 (1) | 0 (0)
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urine color change (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Participants Who Did Not Receive rhIL-7 (N=6) | Arm B - Participants Who Received rhIL-7 (N=26)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 (3) | 8 (16)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (3) | 9 (18)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 10 (20)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (4) | 5 (9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 3 (3)
Allergy/Immunology - Other (runny nose/allergy) (Immune system disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 4 (4)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (fast heartbeat) (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac General - Other (tachycardia) (Cardiac disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constitutional Symptoms - Other (weakness) (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Dental: teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatology/Skin-Other (dermatitis; eczema; erythema) (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (4) | 6 (8)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 5 (5)
Flu-like syndrome (General disorders) | 0 (0) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 5 (9)
Glucose, serum-high (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 11 (24)
Hemorrhage, GU: Urinary NOS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory: Nose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Injection - Other (upper respiratory infection) (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 4 (12) | 21 (22)
Insomnia (General disorders) | 0 (0) | 1 (1)
Low Leukocytes (total WBC) count (Blood and lymphatic system disorders) | 5 (5) | 8 (23)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5) | 18 (47)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (7) | 9 (17)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (6)
Mood alteration: anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Nasal cavity/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (6)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2) | 11 (25)
Ocular/Visual-Other, (Edema: eye; itching: eye) (Eye disorders) | 1 (2) | 0 (0)
PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain: Other (General disorders) | 2 (2) | 4 (4) — (Inj. site; mouth; Pain: left sacrum and groin area; pain: shoulder; pain:wrist/arms; pain: injection site)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Pain: Buttock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain: External ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain: Head/headache (Nervous system disorders) | 0 (0) | 2 (2)
Pain: joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Phosphate, serum low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
Low Platelets (Blood and lymphatic system disorders) | 1 (1) | 13 (24)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8)
Pulmonary/Upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — Sinus congestion: runny/stuffy nose; wheezing
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rigors/Chills (General disorders) | 1 (1) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Supraventricular & nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (neutralizing antibody) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Re: Reason stopped: Of 30 pts who have received immunotherapy,12 remain on F/U, are stable or without evidence of disease,11 died of PD, 7 are currently receiving additional therapy (NOT ON THIS PROTOCOL) for PD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT00923351/Prot_ICF_000.pdf